CLINICAL TRIAL: NCT00367068
Title: Intrathecal Baclofen. Evaluation of a Therapy for Refractory Spasticity in Children With Cerebral Palsy
Brief Title: Dutch National ITB Study in Children With Cerebral Palsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Medtronic (Industry)
Organization: Maastricht University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF-147
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Cerebral Palsy; Spasticity
Keywords: Cerebral palsy; Spasticity; Child; Baclofen; Intrathecal injection
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Baclofen; Infusion Pumps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: baclofen, intrathecal
Device: infusion pump for intrathecal baclofen, Synchromed, Medtronic

SUMMARY:
The objective of this study is to determine the efficacy and safety of treatment with intrathecal baclofen for severe spasticity in children with cerebral palsy.

DETAILED DESCRIPTION:
Spasticity in cerebral palsy (CP) is a serious problem leading to pain, sleep disturbance, increased expenditure of energy and/or interference with positioning, transfers, dressing and body hygiene. In later stages, secondary phenomena, such as contractures, decubitus and heterotopic calcifications of joints or tendons may create large treatment problems. A substantial group of children with severe CP does not respond to regular treatments, such as physical therapy, orthopaedic surgery or oral medication. An effective treatment option for intractable spasticity is the continuous delivery of intrathecal baclofen (CITB). In 2000, the American Academy for Cerebral Palsy and Developmental Medicine (AACPDM) published a systematic review on the body of evidence about intrathecal baclofen (ITB) for spasticity in individuals with CP. It appeared that only a small and uncertain number of children had been studied. Except for two case-reports, none of the studies solely concerned children. The research methodology employed in three quarters of the available studies was not capable of confirming treatment effect. The AACPDM underlined the need for further high-level research in the form of prospective, randomized trials that use valid and reliable outcome measures in well described and homogeneous groups.

In 1998 the Dutch Study Group on Child Spasticity designed the Dutch national study on the effectiveness and safety of ITB for refractory spasticity in children with cerebral palsy. The Dutch national ITB study included four phases: 1] the selection phase, 2] the double-blind, placebo-controlled dose-escalation test treatment phase, 3] the prospective, randomized, open-label implantation phase and 4] the follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* age between 4 and 16 years
* spastic diplegia or tetraplegia as part of CP
* insufficient response to oral spasticity-reducing medication
* in a mixed CP syndrome, spasticity has to be the most prominent sign
* spasticity results in a decrease in the quality of life of the child and/or its caregivers
* sufficient motivation for participation in the study including availability for follow-up
* magnetic resonance imaging of the brain rules out progressive causes of spasticity

Exclusion Criteria:

* hypersensitivity to baclofen
* contraindications for general anaesthesia
* insufficient general health
* intractable epileptic seizures
* infection of the lumbar skin
* a systemic infection

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18
Dates: Start 2002-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
For the double-blind, placebo-controlled dose-escalation test treatment phase:
original Ashworth Scale.
For the prospective, randomized, open-label implantation and follow-up phase:
PEDI, GMFM, original Ashworth Scale, Visual Analogue Scale (VAS) at 6 months.

SECONDARY OUTCOMES:
For the double-blind, placebo-controlled dose-escalation test treatment phase:
Visual Analogue Scale (VAS).
For the prospective, randomized, open-label implantation and follow-up phase:
CHQ-PF50 at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Johan SH Vles, MD, PhD, Prof, Study Chair — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Background] Butler C, Campbell S. Evidence of the effects of intrathecal baclofen for spastic and dystonic cerebral palsy. AACPDM Treatment Outcomes Committee Review Panel. Dev Med Child Neurol. 2000 Sep;42(9):634-45. doi: 10.1017/s0012162200001183. No abstract available. PMID 11034458